CLINICAL TRIAL: NCT04653389
Title: Perioperative Multidisciplinary Therapy for Technically Resectable Hepatocellular Carcinoma With Vein Thrombosis: An Exploratory Clinical Trail
Brief Title: Perioperative Therapy for Hepatocellular Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The treatment efficacy was not satisfactory.
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CISLD-10
Record Dates: First submitted 2020-11-28; First posted 2020-12-04 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Vein tumor thrombus; Transarterial chemoembolization; Immunotherapy; Radiotherapy; Multi-disciplinary treatment
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — sintilimab; Immunotherapy; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Single Group Assignment A Phase II Single-arm, Open-label Study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preoperative TACE+Sintilimab+/-Radiotherapy of vein tumor thrombus+postoperative Sintilimab (Experimental): The first TACE and immunotherapy will be performed at the same time on the first day of treatment. Anti-PD-1 Injection will be administered every three weeks ,until the disease progresses according to mRECIST criteria or intolerable toxicity or the patients' request, or surgery.Hypofractionated radiation therapy will be adopted for Type Vp2, Vp3 PVTT or Type Vv2 HVTT about 2 weeks after the first TACE.If the imaging examination 4 weeks after the surgery confirm that there is no recurrence and no contraindications to receive immunotherapy, anti-PD-1 antibody adjuvant therapy can be started.Every 21 days is a course of treatment, and the longest medication duration lasts for 6 months.
  Interventions: Drug: Sintilimab Injection; Drug: TACE; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Sintilimab Injection — Sintilimab Injection is used as neoadjuvant therapy and adjuvant therapy.
  Other Names: Immunotherapy; Anti-PD-1 therapy
Drug: TACE — The first TACE and Sintilimab Injection will be initiated simultaneously.
  Other Names: Transarterial Chemoembolization
Radiation: Radiotherapy — Use Cone Beam computor tomography(CBCT) locates the lession before the therapy.
  Other Names: hypofractionated radiation therapy

SUMMARY:
This study aims to observe and evaluate the efficacy and safety of the perioperative multidisciplinary therapy that combines the preoperative transarterial chemoembolization(TACE) and the anti-programmed-death-1 antibody (anti-PD-1) Sintilimab Injection with or without radiotherapy of vein tumor thrombus followed by postoperative anti-PD-1 injection in the treatment of technically resectable hepatocellular carcinoma patients with vein thrombosis.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) has an insidious onset, high degree of invasion, and rapid disease progression. Tumor cells can easily invade the intrahepatic vasculature, especially the portal vein or hepatic venous system, and form portal vein tumor thrombus (PVTT) or hepatic vein tumor thrombus (HVTT).PVTT/HVTT is one of the main adverse factors for the long-term survival of HCC. The location and scope of its occurrence are closely related to the prognosis, and it is also a main hindrance to the improvement of the overall curative effect of HCC in recent years.

As the treatment of HCC converts to multi-disciplinary therapy, the neoadjuvant therapy will be commonly used in the treatment of HCC with PVTT.Early clinical data already support a safe combination of immune checkpoint inhibition with TACE. Moreover，The preliminary results of our previous trial (CISLD-5) showed that TACE combined with anti-programmed-death-1 antibody in patients with BCLC stage A/B HCC beyond Milan criteria has a significant effect.In addition, radiation therapy (RT) can irradiate both the tumor thrombus and the primary tumor .In numbers of retrospective studies, preoperative radiotherapy can achieve radical resection in some patients.

This study is to analyze the safety and efficacy of preoperative TACE and anti-PD-1 Injection combined with or without preoperative radiotherapy of vein tumor thrombus and postoperative anti-PD-1 injection in the treatment of technically resectable hepatocellular carcinoma patients with vein thrombosis.

ELIGIBILITY:
Inclusion Criteria:

1. Newly histologically confirmed diagnosis of HCC or strictly consistent with the clinical diagnostic criteria for HCC according to AASLD guideline；
2. At least one measurable site of disease as defined by modified RECIST (mRECIST) criteria with spiral CT scan or MRI and has not received local treatment；
3. Technically resectable hepatocellular carcinoma with ipsilateral vein tumor thrombosis, including Vp1, Vp2, Vp3 portal vein tumor thrombus (PVTT) (Japan JSH classification) and/or Vv1, Vv2 hepatic vein tumor thrombus (HVTT) (Japan JSH) Type), but not accompanied with extrahepatic organ metastasis, or main portal vein,contralateral portal vein, superior mesenteric vein, vena cava tumor thrombus.Bile duct tumor thrombus can be allowed;
4. tumor burden below 50% of standard liver volume；
5. ECOG PS score: 0~1 points
6. Child-Pugh A or B (<=7)；
7. Life expectancy of at least 3 months;
8. Subjects with chronic HBV infection must be on antiviral therapy per regional standard of care guidelines prior to initiation of study therapy；
9. Adequate blood count, liver-enzymes, and renal function: laboratory test values meet the following requirements within 7 days prior to enrollment (no blood components, cell growth factors, albumin and other corrective therapy drugs are allowed within 14 days prior to laboratory test):

   1. absolute neutrophil count, ANC≥1.5×10^9/L, platelet, PLT≥80×10^9/L, hemoglobin, HGB≥8.5 g/dL;
   2. total bilirubin, TBIL≤1.5×ULN, alanine aminotransferase, ALT and aspartate transferase, AST≤5×ULN, serum Alb≥28 g/L；
   3. creatinine, Cr ≤ 1.5×ULN or clearance of creatinine, CCr≥ 50mL/min, Urine protein<2+;
   4. INR≤ 2 and APTT≤ 1.5×ULN.
10. Female patients with reproductive potential must have a negative urine or serum pregnancy test within 7 days prior to start of trial；
11. Patients agreed to join the clinical trial and signed informed consent and are willing and able to comply with the protocol for the duration of the study including undergoing treatment, adherence to contraceptive measures, scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Have received local or systemic treatments in the past, including but not limited to TACE, immunotherapy, targeted therapy, radiotherapy, radiofrequency therapy, etc.;
2. Diffuse HCC or accompanied by distant metastasis;
3. fibrolamellar carcinoma of liver,cholangiocarcinoma and mixed liver cancer;
4. Insufficient residual liver volume(According to imaging calculations, if there is no background of cirrhosis, the remaining liver volume is less than 35% of the standard liver volume; if there is a background of cirrhosis, the remaining liver volume is less than 40% of the standard liver volume)
5. Active tuberculosis (TB), who are receiving anti-TB treatment or who received anti-TB treatment within 1 year prior to the first study；Patients with previous or current objective evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, and severe impairment of lung function.
6. Patients With II-IV myocardial ischemia and myocardial infarction, poor control of cardiac arrhythmias; Patients with hypertension who cannot be reduced to the normal range after antihypertensive medication (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg).
7. A history of gastrointestinal perforations and/or fistulas, intestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), inflammatory bowel disease or extensive bowel resection (partial colectomy or extensive small bowel resection with chronic diarrhea), Crohn's disease, ulcerative colitis, or chronic diarrhea within 6 months; Patients with a history of gastrointestinal bleeding or a clear gastrointestinal bleeding tendency in the past 6 months, such as esophageal varices with bleeding risk, local active ulcer lesions, and fecal occult blood (++).
8. Severe bleeding tendency or coagulation dysfunction, or receiving thrombolytic treatment; Any life-threatening bleeding event that has occurred within the previous 6 months, including the need for blood transfusion, surgery or topical treatment, and continued medication.
9. Autoimmune disease requiring systematic treatment or a history of the disease within 2 years. (such as vitiligo, psoriasis, hair loss or graves' disease).
10. Patients with central nervous system diseases (such as primary brain tumors, stroke, epilepsy, etc.) or central nervous system metastasis or known brain metastasis.
11. Acute or chronic active hepatitis B or C infection; Human immunodeficiency virus (HIV) infection (HIV 1/2 antibody positive); . A severe infection that is active or clinically poorly controlled. Severe infections, including but not limited to hospitalization for infection, bacteremia, or complications of severe pneumonia, occurred 1 month before the first study.
12. Contains fibroblastic layer hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, bile duct carcinoma and other components; Other malignancies were diagnosed within 5 years prior to the first administration, excluding radical basal cell carcinoma of the skin, skin squamous cell carcinoma and/or radical resection of carcinoma in situ. If other malignancies or liver cancer are diagnosed more than 5 years before administration, a pathological or cytological diagnosis of the relapsed and metastatic lesions is required.
13. Previous major surgery (craniotomy, thoracotomy, or laparotomy) within 1 month or unhealed wounds, ulcers, or fractures; Severe arteriovenous fistula; Uncontrolled metabolic disorders or other non-malignant organ or systemic disease or cancer secondary reactions and may result in higher medical risk and/or uncertainty in survival evaluation.
14. Treated with immunosuppressive drugs, live attenuated vaccine, systemic immunostimulant therapy, or any anti-PD-1, anti-PD-L1/L2 antibody or other immunotherapy and experimental drugs within 4 weeks or planned during the study period.
15. Other acute or chronic conditions, psychiatric disorders, or laboratory abnormalities that may increase the risk of study participation or administration of the study drug, or interfere with the interpretation of the study results, and classify patients as ineligible to participate in the study at the discretion of the investigator.
16. Patients with a history of hepatic encephalopathy or a history of liver transplantation or patients preparing for liver transplantation;
17. Pregnant or lactating women; Known to be allergic to any antibody-targeted drug or small-molecular-targeted drug ingredient; Or have a history of severe allergic reactions to other monoclonal antibodies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-12-26 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Event Free Survival（EFS） | Observation period 48 months
  The time from the patient received treatment to the disease progressed, or the disease recurred after surgical resection without preoperative disease progression, or died from any cause.

SECONDARY OUTCOMES:
Duration of Response（DOR） | 48 months
  Time between the date of first radiographic documented objective response according to mRECIST for HCC and the date of the radiographic disease progression.
Major Pathological response rate（MPR） | 48 months
  Number of participants experiencing the percentage of the non-viable cancer cells (necrotized or fibrotized) out of the surface expression of the total tumor area is <10%
Disease Free Survival（DFS） | 48 months
  The time from the patient received surgery to the disease progressed, or died from any cause.
Overall survival (OS) | 48 months
  Time from first treatment until death
Adverse events | 48 months
  Safety evaluation was done continuously during treatment by using CTCAE 5.0
Tumor biomarker | 48 months
  Including but not limited to AFP,PD-L1,TMB,MSI,HLA,etc.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No